CLINICAL TRIAL: NCT03145766
Title: Immunogenicity and Safety of a Purified Vero Rabies Vaccine - Serum Free When Administered According to a Simulated Rabies Post-exposure Regimen in Healthy Adults
Brief Title: Immunogenicity and Safety of a Purified Vero Rabies Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VRV11; U1111-1174-4976 (Other: UTN)
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Results first posted 2021-01-28 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Rabies Virus
Keywords: Rabies virus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: VRVg-2 Formulation 1 (Experimental): VRVg-2 formulation 1, intramuscular (IM) injection on Days 0, 3, 7, 14 and 28. Concomitant administration of human rabies immunoglobulins (HRIG) on Day 0.
  Interventions: Biological: VRVg 2; Biological: Human Rabies Immunoglobulins (HRIG)
- Group 2: VRVg-2 Formulation 2 (Experimental): VRVg-2 formulation 2, IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
  Interventions: Biological: VRVg 2; Biological: Human Rabies Immunoglobulins (HRIG)
- Group 3: VRVg-2 Formulation 3 (Experimental): VRVg-2 formulation 3, IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
  Interventions: Biological: VRVg 2; Biological: Human Rabies Immunoglobulins (HRIG)
- Group 4: VRVg-1 (Experimental): VRVg-1 initial formulation, IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
  Interventions: Biological: VRVg 1; Biological: Human Rabies Immunoglobulins (HRIG)
- Group 5: Imovax Rabies (Active Comparator): Imovax Rabies, IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
  Interventions: Biological: Imovax Rabies; Biological: Human Rabies Immunoglobulins (HRIG)

INTERVENTIONS:
Biological: VRVg 2 — Modified formulation 1 (Low) of Purified Vero Rabies Vaccine Serum Free
  Arms: Group 1: VRVg-2 Formulation 1
Biological: VRVg 1 — Initial formulation of Purified Vero Rabies Vaccine Serum Free
  Arms: Group 4: VRVg-1
Biological: Imovax Rabies — Purified inactivated rabies vaccine prepared on human diploid cell cultures
  Arms: Group 5: Imovax Rabies
Biological: VRVg 2 — Modified formulation 2 (Medium) of Purified Vero Rabies Vaccine Serum Free
  Arms: Group 2: VRVg-2 Formulation 2
Biological: VRVg 2 — Modified formulation 3 (High) of Purified Vero Rabies Vaccine Serum Free
  Arms: Group 3: VRVg-2 Formulation 3
Biological: Human Rabies Immunoglobulins (HRIG) — Commercialized formulation of HRIG

SUMMARY:
This multicenter, observer-blind, controlled, randomized, Phase II study was designed to evaluate different formulations of the Purified Vero Rabies Cell vaccine VRVg.

DETAILED DESCRIPTION:
This study assessed different formulations of the modified formulation of VRVg (VRVg 2- formulations 1 [low], 2 [medium] and 3 [high]) tested in parallel to the initial VRVg formulation (VRVg-1) and Imovax Rabies. Immune responses were assessed at Day 14, Day 28, Day 42, and at Month 7. Safety events were also reported.

ELIGIBILITY:
Inclusion Criteria:

An individual must fulfill all of the following criteria in order to be eligible for trial enrollment:

1. Aged 18 to less than 65 years on the day of inclusion.
2. Informed consent form had been signed and dated.
3. Able to attend all scheduled visits and to complied with all trial procedures.
4. Body Mass Index (BMI): 18.5 kilograms per meter square (Kg/m^2) less than or equal to (<=) BMI <= 30 Kg/m^2.

Exclusion Criteria:

An individual fulfilling any of the following criteria was to be excluded from trial enrollment:

1. Participant was pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.
2. Participation at the time of study enrollment or, planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
3. Receipt of any vaccine in the 4 weeks (28 days) preceding the first trial vaccination or planned receipt of any vaccine prior to Visit 6.
4. Previous vaccination against rabies (in pre- or post-exposure regimen) with either the trial vaccine or another vaccine.
5. Receipt of immune globulins, blood or blood-derived products in the past 3 months.
6. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
7. At high risk for rabies infection during the trial (e.g., veterinarians and staff, animal handlers, rabies researchers, or any others whose activities may bring them into frequent contact with rabies virus or animals who had the rabies virus).
8. Known systemic hypersensitivity to any of the vaccine or human rabies immunoglobulins (HRIG) components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
9. Self-reported thrombocytopenia, contraindicating IM vaccination.
10. Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
11. Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
12. Current alcohol abuse or drug addiction.
13. Chronic illness that, in the opinion of the investigator, was at a stage where it might interfere with trial conduct or completion (e.g., cardiac disorders, renal disorders, auto immune disorders, diabetes, psychiatric disorders or chronic infection).
14. Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature greater than or equal to [>=] 100.4 Fahrenheit >=38.0 Celsius). A prospective participant should not be included in the study until the condition had resolved or the febrile event had subsided.
15. Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
16. History of Guillain-Barré syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Investigational Site, Redding, California
  - Investigational Site, San Diego, California
  - Investigational Site, South Miami, Florida
  - Investigational Site, Omaha, Nebraska
  - Investigational Site, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Pichon S, Guinet-Morlot F, Saleh J, Essink B, Pineda-Pena AC, Moureau A, Petit C, Minutello AM. Safety and immunogenicity of three dose levels of an investigational, highly purified Vero cell rabies vaccine: A randomized, controlled, observer-blinded, Phase II study with a simulated post-exposure regimen in healthy adults. Hum Vaccin Immunother. 2023 Dec 15;19(3):2275453. doi: 10.1080/21645515.2023.2275453. Epub 2023 Nov 3. PMID 37921410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 centers in the United States from 17 April 2017 to 08 January 2018.
Pre-assignment Details: A total of 320 participants were enrolled and vaccinated in the study.
Groups:
- Group 1: VRVg-2 Formulation 1: VRVg-2 formulation 1 (Low), intramuscular (IM) injection on Days 0, 3, 7, 14 and 28. Concomitant administration of human rabies immunoglobulins (HRIG) on Day 0.
- Group 2:VRVg-2 Formulation 2: VRVg-2 formulation 2 (Medium), IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
- Group 3: VRVg-2 Formulation 3: VRVg-2 formulation 3 (High), IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
Period: Active Vaccination Phase (Day 0-Day 56)
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Started (Randomized.) | 80 | 80 | 80 | 40 | 40
Vaccination 1 | 80 | 80 | 80 | 39 (1 participant of this arm received Imovax Rabies, and counted in Group 5 for safety analysis.) | 41 (1 participant of Group 4 received Imovax Rabies, and counted in Group 5 for safety analysis.)
Vaccination 2 | 77 (1 participant received Group 2 vaccine: counted in Group 2 for post-vaccination 2 safety analysis.) | 81 (1 participant of Group 1 received Group 2 vaccine: counted in Group 2 for post-vaccination 2 safety.) | 80 | 39 | 39
Vaccination 3 | 78 | 79 | 80 | 39 | 38
Vaccination 4 | 78 | 79 | 80 | 38 | 38
Vaccination 5 | 75 | 78 | 79 | 34 | 37
Completed | 74 | 77 | 78 | 33 | 37
Not Completed | 6 | 3 | 2 | 7 | 3
Not completed — Other Adverse Event (AE) | 1 | 1 | 0 | 1 | 2
Not completed — Non-compliance with the Protocol | 0 | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 3 | 0
Not completed — Voluntary Withdrawal Not Due AE | 4 | 1 | 1 | 1 | 0
Period: Follow-up Phase (Day 56 Till Month 7)
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Started | 74 | 77 | 78 | 33 | 37
Completed | 67 | 75 | 73 | 30 | 34
Not Completed | 7 | 2 | 5 | 3 | 3
Not completed — Non-compliance with the Protocol | 2 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 1 | 4 | 2 | 3
Not completed — Voluntary Withdrawal not due to AE | 1 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: VRVg-2 Formulation 1: VRVg-2 formulation 1 (Low), IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
- Total: Total of all reporting groups
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies | Total
Number analyzed (Participants) | 80 | 80 | 80 | 40 | 40 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (13.4) | 42.6 (13.0) | 41.1 (14.4) | 41.1 (13.5) | 38.9 (13.1) | 41.4 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 35 | 41 | 16 | 22 | 158
  Male | 36 | 45 | 39 | 24 | 18 | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 0 | 1 | 1 | 6
  Asian | 1 | 2 | 3 | 0 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 18 | 18 | 22 | 13 | 7 | 78
  White | 56 | 54 | 55 | 24 | 28 | 217
  More than one race | 2 | 3 | 0 | 1 | 2 | 8
  Unknown or Not Reported | 1 | 1 | 0 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Rabies Virus Neutralizing Antibody (RVNA) Geometric Mean Titers (GMTs) Against Rabies Virus at Day 0
Description: RVNA GMT against rabies virus was assessed using the rapid fluorescent focus inhibition test (RFFIT) assay method.
Time Frame: Day 0
Population: Per-Protocol Analysis Set (PPAS): participants who received at least one dose of the study vaccine without protocol deviations before Day 14 (i.e., 7 days after the 3rd vaccine injection).
Measure: Geometric Mean (95% Confidence Interval); unit: international units per milliliter
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 72 | 75 | 71 | 35 | 34
international units per milliliter | 0.101 [0.099 to 0.102] | 0.100 [NA to NA] — Upper and lower limit of 95% confidence interval (CI) was not estimable because all the participants had same value and no variability was observed. | 0.102 [0.099 to 0.104] | 0.101 [0.099 to 0.103] | 0.100 [NA to NA] — Upper and lower limit of 95% CI was not estimable because all the participants had same value and no variability was observed.

2. Primary Outcome: Rabies Virus Neutralizing Antibody Geometric Mean Titers Against Rabies Virus at Day 14
Description: RVNA GMT against rabies virus was assessed using the RFFIT assay method.
Time Frame: Day 14
Population: Analysis was performed on PPAS.
Measure: Geometric Mean (95% Confidence Interval); unit: international units per milliliter
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 72 | 75 | 71 | 35 | 34
international units per milliliter | 1.28 [0.944 to 1.73] | 1.79 [1.33 to 2.41] | 2.52 [1.93 to 3.28] | 1.38 [0.936 to 2.05] | 1.56 [1.06 to 2.29]

3. Primary Outcome: Rabies Virus Neutralizing Antibody Geometric Mean Titers Against Rabies Virus at Day 28
Description: RVNA GMT against rabies virus was assessed using the RFFIT assay method.
Time Frame: Day 28
Population: Analysis was performed on PPAS. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: international units per milliliter
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 66 | 73 | 68 | 29 | 33
international units per milliliter | 3.22 [2.48 to 4.17] | 4.64 [3.53 to 6.10] | 6.81 [5.52 to 8.39] | 3.04 [1.86 to 4.95] | 4.86 [3.56 to 6.65]

4. Primary Outcome: Rabies Virus Neutralizing Antibody Geometric Mean Titers Against Rabies Virus at Day 42
Description: RVNA GMT against rabies virus was assessed using the RFFIT assay method.
Time Frame: Day 42
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: international units per milliliter
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 69 | 72 | 65 | 30 | 31
international units per milliliter | 8.14 [6.60 to 10.0] | 9.68 [7.50 to 12.5] | 15.6 [12.7 to 19.1] | 6.98 [4.69 to 10.4] | 8.99 [6.48 to 12.5]

5. Primary Outcome: Rabies Virus Neutralizing Antibody Geometric Mean Titers Against Rabies Virus at Month 7
Description: RVNA GMT against rabies virus was assessed using the RFFIT assay method.
Time Frame: Month 7
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: international units per milliliter
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 61 | 71 | 64 | 27 | 31
international units per milliliter | 0.894 [0.667 to 1.20] | 0.971 [0.768 to 1.23] | 1.58 [1.28 to 1.94] | 0.939 [0.634 to 1.39] | 1.01 [0.649 to 1.58]

6. Primary Outcome: Percentage of Participants With Rabies Virus Neutralizing Antibody Titer Greater Than or Equal to (>=) 0.2 IU/mL and >=0.5 IU/mL at Day 0
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. Participants with RVNA titer >=0.2 IU/mL were considered as seropositive.
Time Frame: Day 0
Population: Analysis was performed on PPAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 72 | 75 | 71 | 35 | 34
percentage of participants
  RVNA titer >= 0.2 IU/mL | 0 [0 to 5.0] | 0 [0 to 4.8] | 0 [0 to 5.1] | 0 [0 to 10.0] | 0 [0 to 10.3]
  RVNA titer >= 0.5 IU/mL | 0 [0 to 5.0] | 0 [0 to 4.8] | 0 [0 to 5.1] | 0 [0 to 10.0] | 0 [0 to 10.3]

7. Primary Outcome: Percentage of Participants With Rabies Virus Neutralizing Antibody Titers >=0.2 IU/mL and >=0.5 IU/mL at Day 14
Description: as for outcome 6
Time Frame: Day 14
Population: Analysis was performed on PPAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 72 | 75 | 71 | 35 | 34
percentage of participants
  RVNA titer >= 0.2 IU/mL | 93.1 [84.5 to 97.7] | 96.0 [88.8 to 99.2] | 97.2 [90.2 to 99.7] | 97.1 [85.1 to 99.9] | 97.1 [84.7 to 99.9]
  RVNA titer >= 0.5 IU/mL | 75.0 [63.4 to 84.5] | 81.3 [70.7 to 89.4] | 90.1 [80.7 to 95.9] | 80.0 [63.1 to 91.6] | 88.2 [72.5 to 96.7]

8. Primary Outcome: Percentage of Participants With RVNA Titers >=0.2 IU/mL and >=0.5 IU/mL at Day 28
Description: as for outcome 6
Time Frame: Day 28
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 66 | 73 | 68 | 29 | 33
percentage of participants
  RVNA titers >= 0.2 IU/mL | 98.5 [91.8 to 100] | 98.6 [92.6 to 100] | 100 [94.7 to 100] | 96.6 [82.2 to 99.9] | 100 [89.4 to 100]
  RVNA titers >= 0.5 IU/mL | 93.9 [85.2 to 98.3] | 95.9 [88.5 to 99.1] | 100 [94.7 to 100] | 86.2 [68.3 to 96.1] | 100 [89.4 to 100]

9. Primary Outcome: Percentage of Participants With RVNA Titers >=0.2 IU/mL and >=0.5 IU/mL at Day 42
Description: as for outcome 6
Time Frame: Day 42
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 69 | 72 | 65 | 30 | 31
percentage of participants
  RVNA titers >= 0.2 IU/mL | 100 [94.8 to 100] | 98.6 [92.5 to 100] | 100 [94.5 to 100] | 96.7 [82.8 to 99.9] | 100 [88.8 to 100]
  RVNA titers >= 0.5 IU/mL | 100 [94.8 to 100] | 98.6 [92.5 to 100] | 100 [94.5 to 100] | 96.7 [82.8 to 99.9] | 100 [88.8 to 100]

10. Primary Outcome: Percentage of Participants With RVNA Titers >=0.2 IU/mL and >=0.5 IU/mL at Month 7
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. Participants with RVNA titer >= 0.2 IU/mL were considered as seropositive.
Time Frame: Month 7
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 61 | 71 | 64 | 27 | 31
percentage of participants
  RVNA titers >= 0.2 IU/mL | 93.4 [84.1 to 98.2] | 93.0 [84.3 to 97.7] | 100 [94.4 to 100] | 92.6 [75.7 to 99.1] | 87.1 [70.2 to 96.4]
  RVNA titers >= 0.5 IU/mL | 70.5 [57.4 to 81.5] | 77.5 [66.0 to 86.5] | 92.2 [82.7 to 97.4] | 74.1 [53.7 to 88.9] | 74.2 [55.4 to 88.1]

11. Primary Outcome: Geometric Mean Titer Ratio (GMTR) of Rabies Virus Neutralizing Antibody 7 Days Following Vaccination 3 (Day 14/Day 0)
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs 7 days post 3rd vaccination (i.e., on Day 14) and pre-vaccination on Day 0.
Time Frame: Day 0 (pre-dose) and Day 14 (7 days post-dose 3)
Population: Analysis was performed on PPAS.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 72 | 75 | 71 | 35 | 34
ratio | 12.7 [9.37 to 17.1] | 17.9 [13.3 to 24.1] | 24.8 [19.0 to 32.3] | 13.7 [9.27 to 20.3] | 15.6 [10.6 to 22.9]

12. Primary Outcome: Geometric Mean Titer Ratio of Rabies Virus Neutralizing Antibody 14 Days Following Vaccination 4 (Day 28/Day 0)
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs 14 days post 4th vaccination (i.e., on Day 28) and pre-vaccination on Day 0.
Time Frame: Day 0 (pre-dose) and Day 28 (14 days post-dose 4)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 66 | 73 | 68 | 29 | 33
ratio | 31.9 [24.6 to 41.3] | 46.4 [35.3 to 61.0] | 67.0 [54.4 to 82.6] | 30.0 [18.5 to 48.7] | 48.6 [35.6 to 66.5]

13. Primary Outcome: Geometric Mean Titer Ratio of Rabies Virus Neutralizing Antibody 14 Days Following Vaccination 5 (Day 42/Day 0)
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs 14 days post 5th vaccination (i.e., on Day 42) and pre-vaccination on Day 0.
Time Frame: Day 0 (Pre-dose) and Day 42 (14 days Post-dose 5)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 69 | 72 | 65 | 30 | 31
ratio | 80.7 [65.6 to 99.3] | 96.8 [75.0 to 125] | 153 [125 to 188] | 69.0 [46.4 to 103] | 89.9 [64.8 to 125]

14. Primary Outcome: Geometric Mean Titer Ratio of Rabies Virus Neutralizing Antibody 6 Months Following Last Vaccination (Month 7/Day 0)
Description: RVNA titer against rabies virus was assessed using the RFFIT assay method. GMTRs were calculated as the ratio of GMTs 6 month post last vaccination on Month 7 and pre-vaccination on Day 0.
Time Frame: Day 0 (Pre-dose) and Month 7 (6 Months Post Last Vaccination)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 61 | 71 | 64 | 27 | 31
ratio | 8.86 [6.66 to 11.8] | 9.71 [7.68 to 12.3] | 15.5 [12.6 to 19.0] | 9.27 [6.26 to 13.7] | 10.1 [6.49 to 15.8]

15. Primary Outcome: Percentage of Participants With Complete Virus Neutralization at Starting Dilution (1/5) of Rapid Fluorescent Focus Inhibition Test Assay at Day 0
Description: Complete virus neutralization was defined as absence of fluorescent cells at the participant/time point level at the starting dilution (1/5) of the RFFIT assay. Percentage of participants with complete virus neutralization were reported.
Time Frame: Day 0
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 72 | 75 | 71 | 34 | 34
percentage of participants | 0 [0 to 5.0] | 0 [0 to 4.8] | 0 [0 to 5.1] | 0 [0 to 10.3] | 0 [0 to 10.3]

16. Primary Outcome: Percentage of Participants With Complete Virus Neutralization at Starting Dilution (1/5) of Rapid Fluorescent Focus Inhibition Test Assay at Day 14
Description: as for outcome 15
Time Frame: Day 14
Population: Analysis was performed on PPAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 72 | 75 | 71 | 35 | 34
percentage of participants | 79.2 [68.0 to 87.8] | 89.3 [80.1 to 95.3] | 93.0 [84.3 to 97.7] | 82.9 [66.4 to 93.4] | 85.3 [68.9 to 95.0]

17. Primary Outcome: Percentage of Participants With Complete Virus Neutralization at Starting Dilution (1/5) of Rapid Fluorescent Focus Inhibition Test Assay at Day 28
Description: as for outcome 15
Time Frame: Day 28
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 69 | 74 | 70 | 32 | 33
percentage of participants | 92.8 [83.9 to 97.6] | 94.6 [86.7 to 98.5] | 98.6 [92.3 to 100] | 100 [89.1 to 100] | 93.9 [79.8 to 99.3]

18. Primary Outcome: Percentage of Participants With Complete Virus Neutralization at Starting Dilution (1/5) of Rapid Fluorescent Focus Inhibition Test Assay at Day 42
Description: as for outcome 15
Time Frame: Day 42
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 69 | 74 | 68 | 31 | 33
percentage of participants | 97.1 [89.9 to 99.6] | 93.2 [84.9 to 97.8] | 94.1 [85.6 to 98.4] | 100 [88.8 to 100] | 93.9 [79.8 to 99.3]

19. Primary Outcome: Percentage of Participants With Complete Virus Neutralization at Starting Dilution (1/5) of Rapid Fluorescent Focus Inhibition Test Assay at Month 7
Description: as for outcome 15
Time Frame: Month 7
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 61 | 71 | 65 | 27 | 31
percentage of participants | 95.1 [86.3 to 99.0] | 88.7 [79.0 to 95.0] | 100 [94.5 to 100] | 85.2 [66.3 to 95.8] | 93.5 [78.6 to 99.2]

20. Primary Outcome: Number of Participants With Immediate Unsolicited Adverse Events
Description: An adverse event was defined as any untoward medical occurrence in a participant who received study drug and does not necessary have to have a causal relationship with treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report form (CRF) in terms of diagnosis and/or onset post-vaccination. All participants were observed for 30 minutes after any vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRF. Immediate AEs considered as related to vaccination were recorded as immediate unsolicited adverse reactions (ARs).
Time Frame: Within 30 Minutes After any Vaccination
Population: Analysis was performed on safety analysis set (SafAS) that included participant who had received at least one least one dose of the study vaccine and were analyzed according to the actual treatment received. 1 participant of Group 4 received Imovax Rabies, and thus counted in Group 5 for safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 80 | 80 | 80 | 39 | 41
Participants
  Immediate Unsolicited AE | 0 | 1 | 0 | 0 | 2
  Immediate Unsolicited AR | 0 | 1 | 0 | 0 | 2

21. Primary Outcome: Number of Participants With at Least One Solicited Injection Site Reactions
Description: A solicited reaction (SR) was an AR observed and reported under conditions (symptoms and onset) prelisted (i.e., solicited) in the CRF and considered as related to vaccination. An AR was all noxious and unintended responses to a medicinal product related to any dose. Solicited injection site reactions included pain, erythema and swelling at and around the injection site.
Time Frame: Within 7 Days After any and each vaccination (Vaccination 1, 2, 3, 4 and 5)
Population: Analysis performed on SafAS. Here, 'number analyzed' = participants with available data for each specified category.1 participant of Group 4 received Imovax Rabies, and thus counted in Group 5 for safety analysis. At Vaccination 2, 1 participant of Group 1 received Group 2 vaccine and thus counted in Group 2 for post-vaccination 2 safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 80 | 81 | 80 | 39 | 41
Participants
  Pain post-any vaccination: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Pain post-any vaccination | 29 | 32 | 38 | 14 | 24
  Pain Post-vaccination 1: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Pain Post-vaccination 1 | 13 | 20 | 26 | 10 | 16
  Pain Post-vaccination 2: number analyzed (Participants) | 77 | 81 | 80 | 39 | 38
  Pain Post-vaccination 2 | 12 | 12 | 18 | 6 | 10
  Pain Post-vaccination 3: number analyzed (Participants) | 77 | 79 | 80 | 38 | 37
  Pain Post-vaccination 3 | 14 | 10 | 20 | 4 | 9
  Pain Post-vaccination 4: number analyzed (Participants) | 76 | 77 | 80 | 36 | 37
  Pain Post-vaccination 4 | 16 | 11 | 17 | 6 | 11
  Pain Post-vaccination 5: number analyzed (Participants) | 73 | 78 | 78 | 34 | 36
  Pain Post-vaccination 5 | 14 | 7 | 14 | 4 | 10
  Erythema post-any vaccination: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Erythema post-any vaccination | 2 | 1 | 3 | 1 | 2
  Erythema Post-vaccination 1: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Erythema Post-vaccination 1 | 0 | 0 | 1 | 1 | 0
  Erythema Post-vaccination 2: number analyzed (Participants) | 77 | 81 | 80 | 39 | 38
  Erythema Post-vaccination 2 | 0 | 0 | 1 | 0 | 0
  Erythema Post-vaccination 3: number analyzed (Participants) | 77 | 79 | 80 | 38 | 37
  Erythema Post-vaccination 3 | 0 | 0 | 0 | 0 | 0
  Erythema Post-vaccination 4: number analyzed (Participants) | 76 | 77 | 80 | 36 | 37
  Erythema Post-vaccination 4 | 2 | 1 | 2 | 0 | 1
  Erythema Post-vaccination 5: number analyzed (Participants) | 73 | 78 | 78 | 34 | 36
  Erythema Post-vaccination 5 | 0 | 1 | 0 | 0 | 1
  Swelling post-any vaccination: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Swelling post-any vaccination | 0 | 1 | 1 | 1 | 2
  Swelling Post-vaccination 1: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Swelling Post-vaccination 1 | 0 | 1 | 0 | 1 | 0
  Swelling Post-vaccination 2: number analyzed (Participants) | 77 | 81 | 80 | 39 | 38
  Swelling Post-vaccination 2 | 0 | 0 | 0 | 0 | 0
  Swelling Post-vaccination 3: number analyzed (Participants) | 77 | 79 | 80 | 38 | 37
  Swelling Post-vaccination 3 | 0 | 0 | 0 | 0 | 0
  Swelling Post-vaccination 4: number analyzed (Participants) | 76 | 77 | 80 | 36 | 37
  Swelling Post-vaccination 4 | 0 | 0 | 1 | 0 | 1
  Swelling Post-vaccination 5: number analyzed (Participants) | 73 | 78 | 77 | 34 | 36
  Swelling Post-vaccination 5 | 0 | 0 | 0 | 0 | 1

22. Primary Outcome: Number of Participants With at Least One Solicited Systemic Reactions
Description: A solicited reaction was an AR observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the CRF and considered as related to vaccination. An AR was all noxious and unintended responses to a medicinal product related to any dose. Solicited systemic reactions included fever, headache, malaise and myalgia.
Time Frame: Within 7 Days After any and each vaccination (Vaccination 1, 2, 3, 4 and 5)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 80 | 81 | 80 | 39 | 41
Participants
  Fever Post-any Vaccination: number analyzed (Participants) | 78 | 80 | 80 | 39 | 39
  Fever Post-any Vaccination | 0 | 1 | 2 | 0 | 0
  Fever Post-vaccination 1: number analyzed (Participants) | 77 | 80 | 80 | 39 | 39
  Fever Post-vaccination 1 | 0 | 0 | 0 | 0 | 0
  Fever Post-vaccination 2: number analyzed (Participants) | 77 | 81 | 80 | 39 | 38
  Fever Post-vaccination 2 | 0 | 0 | 0 | 0 | 0
  Fever Post-vaccination 3: number analyzed (Participants) | 77 | 78 | 80 | 37 | 37
  Fever Post-vaccination 3 | 0 | 1 | 2 | 0 | 0
  Fever Post-vaccination 4: number analyzed (Participants) | 76 | 77 | 79 | 36 | 37
  Fever Post-vaccination 4 | 0 | 0 | 0 | 0 | 0
  Fever Post-vaccination 5: number analyzed (Participants) | 73 | 77 | 78 | 32 | 36
  Fever Post-vaccination 5 | 0 | 0 | 0 | 0 | 0
  Headache Post-any Vaccination: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Headache Post-any Vaccination | 26 | 12 | 20 | 9 | 15
  Headache Post-vaccination 1: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Headache Post-vaccination 1 | 11 | 8 | 15 | 5 | 9
  Headache Post-vaccination 2: number analyzed (Participants) | 77 | 81 | 80 | 39 | 38
  Headache Post-vaccination 2 | 11 | 3 | 5 | 1 | 9
  Headache Post-vaccination 3: number analyzed (Participants) | 77 | 79 | 80 | 38 | 37
  Headache Post-vaccination 3 | 14 | 4 | 5 | 2 | 10
  Headache Post-vaccination 4: number analyzed (Participants) | 76 | 77 | 80 | 36 | 37
  Headache Post-vaccination 4 | 6 | 4 | 9 | 3 | 5
  Headache Post-vaccination 5: number analyzed (Participants) | 73 | 78 | 78 | 34 | 36
  Headache Post-vaccination 5 | 7 | 1 | 7 | 1 | 7
  Malaise Post-any Vaccination: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Malaise Post-any Vaccination | 26 | 13 | 17 | 11 | 16
  Malaise Post-vaccination 1: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Malaise Post-vaccination 1 | 14 | 8 | 10 | 6 | 9
  Malaise Post-vaccination 2: number analyzed (Participants) | 77 | 81 | 80 | 39 | 38
  Malaise Post-vaccination 2 | 8 | 3 | 7 | 2 | 10
  Malaise Post-vaccination 3: number analyzed (Participants) | 77 | 79 | 80 | 38 | 37
  Malaise Post-vaccination 3 | 8 | 4 | 3 | 3 | 5
  Malaise Post-vaccination 4: number analyzed (Participants) | 76 | 77 | 80 | 36 | 37
  Malaise Post-vaccination 4 | 6 | 4 | 10 | 6 | 6
  Malaise Post-vaccination 5: number analyzed (Participants) | 73 | 78 | 78 | 34 | 36
  Malaise Post-vaccination 5 | 5 | 1 | 5 | 4 | 4
  Myalgia Post-any Vaccination: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Myalgia Post-any Vaccination | 25 | 22 | 20 | 11 | 19
  Myalgia Post-vaccination 1: number analyzed (Participants) | 79 | 80 | 80 | 39 | 39
  Myalgia Post-vaccination 1 | 16 | 14 | 15 | 5 | 13
  Myalgia Post-vaccination 2: number analyzed (Participants) | 77 | 81 | 80 | 39 | 38
  Myalgia Post-vaccination 2 | 9 | 3 | 6 | 6 | 8
  Myalgia Post-vaccination 3: number analyzed (Participants) | 77 | 79 | 80 | 38 | 37
  Myalgia Post-vaccination 3 | 8 | 7 | 5 | 3 | 9
  Myalgia Post-vaccination 4: number analyzed (Participants) | 76 | 77 | 80 | 36 | 37
  Myalgia Post-vaccination 4 | 9 | 7 | 5 | 4 | 5
  Myalgia Post-vaccination 5: number analyzed (Participants) | 73 | 78 | 78 | 34 | 36
  Myalgia Post-vaccination 5 | 7 | 5 | 10 | 3 | 9

23. Primary Outcome: Number of Participants With at Least One Unsolicited Adverse Events
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and does not necessary have to have a causal relationship with treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the CRF in terms of diagnosis and/or onset post-vaccination.
Time Frame: Within 28 Days After any vaccination
Population: Analysis was performed on SafAS. 1 participant of Group 4 received Imovax Rabies vaccine, and thus counted in Group 5 for safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 80 | 80 | 80 | 39 | 41
Participants | 11 | 11 | 20 | 10 | 18

24. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and does not necessary have to have a causal relationship with treatment. An SAE was any untoward medical occurrence that at any dose resulted in death; life-threatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect or a medically important event.
Time Frame: From Day 0 up to Month 7
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2:VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
Number analyzed (Participants) | 80 | 80 | 80 | 39 | 41
Participants | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data were collected from Day 0 (post-vaccination 1) up to 28 days post any vaccination. SR data were collected within 7 days post any vaccination. SAE data were collected throughout the study (up to 6 months after last vaccination, i.e., up to Month 7).
Description: Analysis was performed on SafAS. A SR was an AE that was prelisted (i.e., solicited) in the CRF and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the CRF in terms of diagnosis and/or onset post-vaccination.
Groups:
- Group 2: VRVg-2 Formulation 2: VRVg-2 formulation 2 (Medium), IM injection on Days 0, 3, 7, 14 and 28. Concomitant administration of HRIG on Day 0.
Arm/Group | Group 1: VRVg-2 Formulation 1 | Group 2: VRVg-2 Formulation 2 | Group 3: VRVg-2 Formulation 3 | Group 4: VRVg-1 | Group 5: Imovax Rabies
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80 | 0/80 | 0/39 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 1/80 | 0/39 | 0/41
Other Adverse Events (participants affected / at risk) | 40/80 | 39/80 | 45/80 | 22/39 | 28/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: VRVg-2 Formulation 1 (N=80) | Group 2: VRVg-2 Formulation 2 (N=80) | Group 3: VRVg-2 Formulation 3 (N=80) | Group 4: VRVg-1 (N=39) | Group 5: Imovax Rabies (N=41)
Facial Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: VRVg-2 Formulation 1 (N=80) | Group 2: VRVg-2 Formulation 2 (N=80) | Group 3: VRVg-2 Formulation 3 (N=80) | Group 4: VRVg-1 (N=39) | Group 5: Imovax Rabies (N=41)
Application Site Bruise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Injection Site Pain (General disorders) | 29 (69) | 32 (60) | 38 (95) | 14 (30) | 24 (56)
Malaise (General disorders) | 26 (41) | 13 (20) | 17 (35) | 11 (21) | 16 (35)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (49) | 22 (36) | 20 (41) | 11 (21) | 19 (44)
Headache (Nervous system disorders) | 26 (49) | 12 (20) | 21 (42) | 10 (13) | 15 (41) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT03145766/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT03145766/SAP_001.pdf